CLINICAL TRIAL: NCT04765293
Title: The Effect of GRAVITY System Therapy on Chronic Low Back Pain in Disc Disease
Brief Title: GRAVITY System Therapy on Chronic Low Back Pain
Acronym: GRAVITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Aleksandra Truszczynska Baszak, Assoc Prof, Józef Piłsudski University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Research Group no 4; SN 4 (Other Grant/Funding Number: Research Group no 4 at Jozef Pilsudski University of Physical Education)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Physical Therapy; Low Back Pain; Chronic Pain
Keywords: gravity system; strengthening exercises; disability
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor was blinded concerning participants therapy model and results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gravity group (Experimental): GRAVITY® system exercise is conducted on a machine. The tasks were non-weight bearing, and the only external load was the body mass of the trainee. The degree of unloading (the level of exercise) was chosen depending on the patient's body mass, their current health and the difficulty of the exercise. The machine allowed for exercising any chosen muscle group at chosen setting of the bench, platform and ropes. GRAVITY® system exercise aimed at general posture improvement and at strengthening the desired movement path, along with strengthening the deep spinal and abdominal muscles.
  GRAVITY therapy group had therapy twice a week for 4 weeks for 40 minutes that made 2x40 minx 4 weeks=320 minutes.
  Interventions: Other: Physical Therapy
- Control group (Active Comparator): Control group had standard, two weeks ambulant every day physical therapy sessions ( laser therapy, cryotherapy, magnetotherpy, TENS and interference currents), 5 times a week 30 min, that is 10 sessions 30 min x10=300 min.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical Therapy Gravity strengthening exercises vs standard physical therapy
  Other Names: Gravity vs standard physical therapy

SUMMARY:
The aim of the study was to examine the effect of GRAVITY system therapy on chronic disc-related pain in lumbar spine. Investigators made a hypothesis that patients who regularly perform core strengthening exercises based on gravity system will decrease pain and disability, and increase muscle strength in higher extent comparing to control group, that receive passive physical therapy.

DETAILED DESCRIPTION:
GRAVITY therapy group had therapy twice a week for 4 weeks for 40 minutes that made 2x40 minx 4 weeks=320 minutes.

Clinical control group had standard, two weeks ambulant, every day, physical therapy sessions, 5 times a week 30 min, that is 10 sessions 30 min x10=300 min. So the total amount of treatment was comparable.

All participants in both groups completed the study. Investigators used the Oswestry Disability Index (ODI) to determine the disability level of patient with low back pain (Shah et al, 2016), and VAS scale (visual analogue scale) (0-10) to measure pain intensity.

The next stage of examination was the lumbopelvic complex stability test. The test comprised of several activities which had to be performed without lifting the lumbar region. The more difficult activity a patient was able to perform, the higher was assessed their muscle strength.

All the patients were examined twice:

1. before starting the therapy cycle,
2. and after the therapy. They were informed about the aim of the study, the study course and the possible risks. The participation in the study was voluntary and anonymous. The patients signed informed consent to participate in the study. The next step was the lumbopelvic complex stability test. Patients took it in lying position. The therapist placed their hand under the patient's lumbar region, with the patient's spinous processes resting on second do fifth metacarpal heads. Then, the therapist instructed the patient on the type of movement the patient was supposed to perform. The patient's task was to perform the task without lifting the lumbar region off the therapists' fingers. If the task was performed correctly, the next level task ensued. If the patient lifted their lumbar region, it meant that they did not have enough muscle strength for that level. The test was to be performed without pain, and if the patient felt pain, the test was discontinued and the patient was assigned muscle strength from the level without pain syndromes. Each correctly performed task translated into a given level of muscle strength.

Level 0.3 - lying on the back with the limbs flexed at the hips and knees. The patient drew the knee to the chest, then returned to the starting position. Level 0.4 - lying on the back, the patient held flexed leg with their arms at their chest, and then drew the other leg. Level 0.5 - the same exercise as in position 0.4, yet without stabilizing the leg with the arms. Level 1a - one leg flexed at the hip and the knee, the other leg was lying extended and then it was raised upwards, extended. Then, the patient swapped legs and repeated the task. Level 1b - patient position as in 1a, yet the extended leg was brought up to the flexed leg. Then the patient swapped legs and repeated the exercise. Level 2 - one leg was flexed at 90° at the hip and at the knee, the other leg was extended. The patient extended the flexed leg, sliding the heel on the ground. After the knee was fully extended, the leg returned to the starting position. Then the patient swapped legs. Level 3 - the patient flexed first one leg and then the other leg to 90°, and then extended first one leg and then the other leg and slid them out on the ground. After the knee was fully extended, the limb returned to the starting position. Level 4 - both legs were extended on the ground, then the patient flexed both limbs sliding their heel on the ground, and then lifted then, flexing the leg at the hip to 90° and returned to starting position. Level 5 - starting position as in level 4, the patient flexed legs at the hip and the knee and drew them to the chest, then the patient extended both legs simultaneously at the hip and the knee, thus returning to the starting position.

Therapy GRAVITY® system exercise is conducted on a machine. The tasks were non-weight bearing, and the only external load was the body mass of the trainee. The degree of unloading (the level of exercise) was chosen depending on the patient's body mass, their current health and the difficulty of the exercise. The machine allowed for exercising any chosen muscle group at chosen setting of the bench, platform and ropes. GRAVITY® system exercise aimed at general posture improvement and at strengthening the desired movement path, along with strengthening the deep spinal and abdominal muscles.

The training sessions started with manometer exercise - the manometer was placed under the lumbar region of the spine. As the patient exhaled and tensed their abdominal muscles, manometer membrane was pumped to 40 mmHg. This provided non-invasive biofeedback, making the patients aware if their deep smooth muscles maintained the desired tension. The patients were to conduct all exercises (knee bends on a sloping bench, lower limb abduction, upper and lower body exercise) while simultaneously maintaining abdominal muscles tension on the level.

Then, the patients conducted their training designed accordingly to their individual needs. The most common exercise set was the following: moving their arms from behind the head in the lying on the back position (2x12 repetitions), abductions to 90° in the lying position (3 sets of 10 repetitions for both the right and the left side), adduction of both arms in the sitting position facing the machine (2x12), pulling the bench (2x12), abdominal oblique muscle tension (2x10) (fig. 2), rotating the trunk in sitting position (2x10 on the right and on the left sides), plank (2x30s), knees to chest (2x10), heels-up on the platform (3x15 left leg, right leg, both feet), steps forward (2x10 right leg and left leg). While exercising, the patients were to maintain the right body posture actively by tensing their abdominal muscles. Each exercise could be performed in several variations, such as: both limbs working out simultaneously, or single limb workout, or increasing the level through making the exercise easier or more difficult to perform. At the end of each training session patients stretched individual muscle groups (e.g. posterior thigh muscles, quadriceps femoris muscle, and triceps surae muscle) or they used rollers.

In the clinical control group, the patients had physical therapy such as: laser therapy, cryotherapy, magnetotherpy, interference currents. They had therapy every day for the period of two weeks.

Both groups had different blinded clinicians supervising therapy. Another specialist collected and analysed the treatment results.

Patients from both groups did not received any other simultaneous treatments (e.g., pharmacological or psychological).

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic, local low back pain
* diagnosed with lumbar spinal disc disease confirmed with medical examination and anamnesis by a physiotherapist/ neurosurgeon; current MRI scan,
* no history of spinal surgery,
* no earlier physiotherapy

Exclusion Criteria:

* other spinal dysfunctions
* history of spinal surgery,
* physiotherapy attendance before the start of the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Visual Analogue Scale (0-10)

SECONDARY OUTCOMES:
Disability | 4 weeks
  Oswestry Disability Index
Abdominal muscle strength | 4 weeks
  lumbopelvic complex stability test by Sahrmann

CONTACTS AND LOCATIONS:
Locations (1):
- Fizjokoncept, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
row results data

REFERENCES:
- [Background] B Amorim A, Simic M, Pappas E, Zadro JR, Carrillo E, Ordonana JR, Ferreira PH. Is occupational or leisure physical activity associated with low back pain? Insights from a cross-sectional study of 1059 participants. Braz J Phys Ther. 2019 May-Jun;23(3):257-265. doi: 10.1016/j.bjpt.2018.06.004. Epub 2018 Jun 28. PMID 31130170
- [Background] Arab AM, Shanbehzadeh S, Rasouli O, Amiri M, Ehsani F. Automatic activity of deep and superficial abdominal muscles during stable and unstable sitting positions in individuals with chronic low back pain. J Bodyw Mov Ther. 2018 Jul;22(3):627-631. doi: 10.1016/j.jbmt.2017.10.009. Epub 2017 Oct 25. PMID 30100288
- [Background] Barr KP, Griggs M, Cadby T. Lumbar stabilization: core concepts and current literature, Part 1. Am J Phys Med Rehabil. 2005 Jun;84(6):473-80. doi: 10.1097/01.phm.0000163709.70471.42. PMID 15905663